CLINICAL TRIAL: NCT06552871
Title: Participatory Research for Suicide Prevention in Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Anne Kirby, Associate Professor, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 00139671; K23MH123934 (NIH)
Record Dates: First submitted 2024-08-07; First posted 2024-08-14 (Actual); Results first posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Autism; Suicide Prevention
Keywords: educational intervention; pilot test
MeSH Terms: conditions — Autistic Disorder; Suicide Prevention

STUDY DESIGN:
Intervention Model Description: Initial pre-post pilot test
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FLAPS intervention (Experimental): Participants receiving FLAPS intervention
  Interventions: Behavioral: Forming Love around Autistic People to Prevent Suicide

INTERVENTIONS:
Behavioral: Forming Love around Autistic People to Prevent Suicide — Four-part virtual educational intervention
  Other Names: FLAPS

SUMMARY:
The goal of this study is to pilot test a new educational intervention for organization members focused on suicide prevention for autistic people. The main questions it aims to answer are:

* Does participating in the intervention increase participants' knowledge, skills, and actions to support suicide prevention for autistic people?
* What feedback do participants have to help improve the intervention?

Participants will:

* engage in a four-part virtual educational intervention
* answer questions via online survey before, after, and 3-months after the intervention
* participate in an optional interview to provide feedback

DETAILED DESCRIPTION:
This study will pilot test a new four-part virtual educational intervention called Forming Love around Autistic People to Prevent Suicide (FLAPS).

Participants will be active members of an organization (e.g., paid employee, volunteer, stakeholder) whose work impacts autistic people. They will participate in four virtual educational sessions led by trained facilitators.

The educational intervention will provide current research evidence and community-informed information about suicide risk and prevention, and engage participants in active discussions to expand their knowledge and skills as well as to promote action planning to support suicide prevention for autistic people in their community.

Participants will provide demographic and descriptive information and complete the Steps Toward Prevention (Autism Community Suicide Prevention) measure at three time-points (Pre-intervention, post-intervention [approximately 2 months after baseline], and 3-months after intervention). The Steps Toward Prevention (Autism Community Suicide Prevention) measure will assess participants' knowledge, skills, and actions to support suicide prevention for autistic people. They will also be provided an option to complete a short interview to provide feedback about the FLAPS intervention.

ELIGIBILITY:
Inclusion Criteria:

* Active member of an organization whose work impacts autistic people
* Age 18+
* Fluent English language to participate in virtual educational intervention

Exclusion Criteria:

* No access to an internet-connected device
* Unable to participate in a virtual educational intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2024-09-05 (Actual); Primary Completion 2025-08-05 (Actual); Study Completion 2025-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne V Kirby, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kirby AV, Bakian AV, Zhang Y, Bilder DA, Keeshin BR, Coon H. A 20-year study of suicide death in a statewide autism population. Autism Res. 2019 Apr;12(4):658-666. doi: 10.1002/aur.2076. Epub 2019 Jan 21. PMID 30663277
- [Background] Wexler L, McEachern D, DiFulvio G, Smith C, Graham LF, Dombrowski K. Creating a Community of Practice to Prevent Suicide Through Multiple Channels: Describing the Theoretical Foundations and Structured Learning of PC CARES. Int Q Community Health Educ. 2016;36(2):115-22. doi: 10.1177/0272684X16630886. Epub 2016 Feb 15. PMID 26880738
- [Background] Wexler L, Rataj S, Ivanich J, Plavin J, Mullany A, Moto R, Kirk T, Goldwater E, Johnson R, Dombrowski K. Community mobilization for rural suicide prevention: Process, learning and behavioral outcomes from Promoting Community Conversations About Research to End Suicide (PC CARES) in Northwest Alaska. Soc Sci Med. 2019 Jul;232:398-407. doi: 10.1016/j.socscimed.2019.05.028. Epub 2019 May 23. PMID 31151026

RESULTS

PARTICIPANT FLOW:
Groups:
- FLAPS: Assigned to the FLAPS intervention
Period: Overall Study
Arm/Group | FLAPS
Started | 51
Completed | 49
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Enrolled participants were all assigned to the FLAPS intervention
Arm/Group | FLAPS
Number analyzed (Participants) | 51
Age, Customized [Count of Participants; unit: Participants] — Age categories (years)
  Participants
    Age: 18-29 years | 8
    Age: 30-39 years | 17
    Age: 40-49 years | 14
    Age: 50-59 years | 8
    Age: 60+ years | 4
Sex/Gender, Customized [Count of Participants; unit: Participants] — Sex
  Participants
    Sex: Male | 8
    Sex: Female | 40
    Sex: Other/Choose not to respond | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 45
  More than one race | 1
  Unknown or Not Reported | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Hispanic ethnicity
  Participants
    Hispanic or Latino | 14
    Not Hispanic or Latino | 35
    Unknown or Not Reported | 2
Organization (anonymized) [Count of Participants; unit: Participants] — Individual participants were members of existing organization groupings based on their employment or volunteer status with the participating organization (organizations anonymized). These groupings are included in analysis because individuals within organizations are not independent, therefore these groupings are captured at baseline. There are no levels or hierarchical descriptions of the organizations. Organization names presented here are randomly assigned letters.
  Participants
    AA | 1
    AB | 2
    AC | 9
    AD | 6
    AE | 4
    BA | 5
    BB | 1
    BC | 2
    BD | 1
    CA | 15
    CB | 5

OUTCOME MEASURES:

1. Primary Outcome: Steps Toward Prevention - Autism Community Suicide Prevention: Knowledge & Capacity
Description: Self-report measure of knowledge, skills, and actions to support suicide prevention for autistic people. This reported data is for the Knowledge & Capacity scale of the Steps Toward Prevention - Autism Community Suicide Prevention measure. This scale inquires about how true eight statements are for the respondent currently on a 5-point scale (Definitely not true - Definitely true). Scores are averaged across the items (1-5 possible range). Higher numbers indicate greater knowledge and capacity for suicide prevention.
Time Frame: Pre-intervention, post-intervention (approximately 2 months after baseline), and 3-months after intervention
Population: When reporting means here, we report only those who completed the measures at each time point. For the multi-level statistical analyses, we applied baseline-observation-carried-forward to have a complete analysis including all participants.
Measure: Mean (Standard Deviation); unit: Scores on a 5-point scale
Arm/Group | FLAPS
Number analyzed (Participants) | 51
Scores on a 5-point scale
  Pre-study data: Knowledge & Capacity | 3.98 (0.53)
  Post-study data: Knowledge & Capacity: number analyzed (Participants) | 34
  Post-study data: Knowledge & Capacity | 4.54 (0.54)
  Follow-up data: Knowledge & Capacity: number analyzed (Participants) | 28
  Follow-up data: Knowledge & Capacity | 4.52 (0.56)
Statistical Analysis 1: Comparison: FLAPS; Applied baseline-observation-carried-forward to evaluate change in Knowledge & Capacity between pre- and post-intervention, accounting for organization membership; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mixed effects GLM Coefficient = 0.35, Standard Error of Mean 0.07

2. Primary Outcome: Steps Toward Prevention - Autism Community Suicide Prevention: Actions
Description: Self-report measure of knowledge, skills, and actions to support suicide prevention for autistic people. This reported data is for the Actions scale of the Steps Toward Prevention - Autism Community Suicide Prevention measure. This inquires about how often the respondent has done twelve types of actions in the past month on a 5-point scale (Never - More than once a week). Scores are averaged across the items (1-5 possible range). Higher numbers indicate greater engagement in actions for suicide prevention.
Time Frame: Pre-intervention, post-intervention (approximately 2 months after baseline), and 3-months after intervention
Population: When reporting means here, we report only those who completed the measures at each time point. For the multi-level statistical analyses, we applied baseline-observation-carried-forward to have a complete analysis including all participants. Baseline data for actions is only available for N=50 because one participant did not complete this section of the baseline questionnaire prior to study start.
Measure: Mean (Standard Deviation); unit: Scores on a 5-point scale
Arm/Group | FLAPS
Number analyzed (Participants) | 50
Scores on a 5-point scale
  Pre-study data: Actions | 2.95 (0.93)
  Post-study data: Actions: number analyzed (Participants) | 34
  Post-study data: Actions | 3.55 (0.83)
  Follow-up data: Actions: number analyzed (Participants) | 28
  Follow-up data: Actions | 3.53 (0.79)
Statistical Analysis 1: Comparison: FLAPS; Applied baseline-observation-carried-forward to evaluate change in Actions between pre- and post-intervention, accounting for organization membership; Test type: Superiority — Applied mixed effects GLM to estimate significant improvement in the outcome measure, while accounting for organization membership (nested participants); p < 0.01, Mixed Models Analysis; Mixed effects GLM Coefficient = 0.38, Standard Error of Mean 0.13

3. Secondary Outcome: Qualitative Interview
Description: Open-ended interview questions to understand additional outcomes that participants experienced that they attribute to the intervention.
Time Frame: Post intervention (approximately 2 months after baseline)
Population: Interviews were optional, not all participants chose to complete one.
Measure: Count of Participants; unit: Participants
Groups:
- Interview Participants: Interviews were optional, only some intervention participants chose to complete an interview after completing FLAPS.
Arm/Group | Interview Participants
Number analyzed (Participants) | 18
Participants
  Enhanced understanding about autism and working with autistic people: Evidence for this theme in interview | 9
  Enhanced understanding about autism and working with autistic people: No evidence for this theme identified | 9
  Enhanced understanding about suicide among autistic people: Evidence for this theme in interview | 17
  Enhanced understanding about suicide among autistic people: No evidence for this theme identified | 1
  Motivation in organization to take steps to reduce suicidality in the autistic population they serve: Evidence for this theme in interview | 18
  Motivation in organization to take steps to reduce suicidality in the autistic population they serve: No evidence for this theme identified | 0

ADVERSE EVENTS:
Time Frame: Not monitored
Description: Not monitored
Groups:
- No Monitoring: Adverse event monitoring did not occur due to low-risk nature of virtual educational intervention.
Arm/Group | No Monitoring
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
We did not measure the long-term effects of the intervention on autistic people and their suicide risk.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-08): https://cdn.clinicaltrials.gov/large-docs/71/NCT06552871/Prot_SAP_000.pdf